CLINICAL TRIAL: NCT04354181
Title: Characterising and Fingerprinting Biomarkers of Urolithiasis: A Case Control Study
Brief Title: Urine Biomarker for Stone Recurrence
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE- 2020.058
Record Dates: First submitted 2020-04-08; First posted 2020-04-21 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — about 100 cc urine will be collected for the measurement of Biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the advent of treating stones with Extracorporeal Shock Wave Lithotripsy (ESWL) and Percutaneous nephrolithotomy (PCNL), the recurrence rate for renal stones remains high and this may be due to poor compliance of patients with dietary and fluid advice, age, metabolic abnormalities, medicines and the formation of "new stones" from clinically insignificant residual fragments (CIRF).

Though some patients become stone-free after ESWL/PCNL or open surgeries, the majority develop "new stones" and it is difficult to predict when these stones will recur until either they have imaging perform or they developed symptoms. However, the use of regular imaging for monitoring will be costly and involve radiation exposure. Therefore, a diagnostic tool is needed to enable the clinician and/or patient to monitor for stone recurrence.

In the previous studies, some urine markers were identified that are related to stone formation. The relationship of these urine markers with the recurrence of renal stone will be further explore in this study. Also, potential markers that could predict stone recurrence will be identified, and hence earlier intervention could be offered to patients.

DETAILED DESCRIPTION:
Stone recurrences remain a major challenge in the management of renal stone patients, despite the emergence of ESWL as an internationally accepted method for the minimally invasive treatment of most renal stones . Depending on the location and size of a stone, the success rates for ESWL can be greater than 80% for successful disintegration (fragmentation) of the stone, and the rate at which patients remain stone-free after 3 months ranges from 40%-80%. The rates of stone recurrence, defined as symptomatic episodes and/or interventions due to residual fragments, after ESWL, PCNL and URETS range from 10%-60% and depend upon the duration of the prospective follow-up study. In long-term follow-up studies after ESWL, the recurrence rates have been shown to increase annually. This recurrence could be due to poor patient compliance with dietary and fluid-intake advice, patient age, metabolic abnormalities, the side-effects of medicines or the formation of new stones from the CIRFs that result from ESWL.

The fragments of clinically insignificant or significant stones that remain after ESWL/PCNL/URETS can pose a long-term risk for patients by serving as a nidus for new stone formation. Patients are declared 'stone-free' after ESWL only if no fragments are detected on radiographs, ultrasound scans or intravenous pyelograms with tomography and spiral computed tomography (CT) scans. Fragments smaller than 5 mm are considered capable of spontaneous passage, and such fragments are regarded as CIRF. Despite prophylactic measures to reduce stone formation, the recurrence rate remains high. There is also a paucity of information concerning the biochemical or metabolic evaluations of patients who have been tracked in the long-term studies described above. Some specific biological effects from ESWL are well known; for example, the urinary enzyme levels are known to increase. Although the enzyme levels commonly return to normal in the short-term, the levels of these enzymes, and other biomarkers such as glycosaminoglycans and cytokines, have not been tracked over longer periods of time.

The urinary levels of both cytokines and mediators of inflammation are becoming increasingly recognised as important markers for urologic diseases. In a study of the urinary levels of IL-6, IL-1β and 1α in patients with stone disease, patients without bacterial cystitis showed significant elevations of IL-6 but did not have marked increases in either IL-1β or 1α relative to control subjects. The patients with bacterial cystitis showed elevations in all three cytokines. Studies have also examined the injury to cells from oxalate toxicity and calcium oxalate crystal exposure, using tests on tissue cultures and rat models [20-22]. Such types of cellular damage have also been shown to attract crystal binding, which can lead to crystal growth and aggregation. An inflammatory response has also been seen in experimental nephrolithiatic rats, whereby crystals were shown to form in the tubular lumen and eventually to move into the interstitium, causing inflammation and attracting macrophages or other inflammatory cells. Recent advances in translational medicine have also identified new molecules such as urinary kidney injury molecule-1 (uKIM-1). The levels of the uKIM-1 molecule have been found to be increased following lithotripsy, suggesting it might be a good candidate for an acute kidney injury (AKI) molecule. Hence, studying the levels of cytokines and the mediators of inflammation could help in understanding the pathogenesis of urolithiasis. Such studies could also identify a reliable marker for the early diagnosis, treatment and prevention of stone recurrence.

Small fragments (<5 mm) that have not passed spontaneously and are retained undetected in the urinary tract can develop into new stones in the ensuing months or years. The investigators hypothesise that such retained fragments are most likely to be attached to the urothelium, thereby injuring the cells and the underlying tissue. The investigators also hypothesise that depending on the growth rate of a fragment, this injury can invoke an inflammatory response that begins as sub-clinical (i.e., asymptomatic). This kind of injury is akin to stone-formation causing mechanical stimulation (i.e., irritation) of the epithelial cells, which results in the production of cytokines and mediators of inflammation. These by-products eventually become a 'plaque', similar to a Randall's plaque. These hypotheses have been recently reviewed and have been suggested to indicate a likely pathway to calcium stone formation.

In previous studies on the separation of urinary glycosaminoglycans (GAGs), the investigators have reported the electrophoretic separation of urinary GAGs into their sub-classes on a preparative scale. Chondroitin sulphates (CS) and HAs were cleanly separated from the heparan sulphates (HS). On further analysis by high-performance liquid chromatography, HAs were identified as the major contributors to the crystallisation-promoting properties observed in the early electrophoretic fractions of stone-formers. The involvement of HAs in urolithiasis was further supported from studies involving their extraction and identification in calcium-containing stones. The investigators also confirmed that the in vivo role of HAs was more likely to be a secondary effect rather than a cause of stone formation, although the release and increase of HAs from injured tissues could accelerate the growth and deposition of calcium and oxalate (e.g., on the CIRF).

In previous preliminary case-controlled study, the investigators had looked into a multitude of potential biomarkers and inflammatory cytokines. The molecular candidates were from both urine and serum samples, and six patient groups were assessed including active stone-formers with and without infection and before and after the removal of stones. Also, normal controls with and without urinary tract infections were assessed.

The most well-studied and characterised markers, which are also easily available, were selected for the study. The markers included: (1) the inflammatory markers IL-1α, IL-6 and IL-8, (2) the mediator macrophage inflammatory protein-1α (MIP-1α) and (3) the urinary biochemical markers N-acetyl-β-D-glucosaminidase (NAG), neutrophil gelatinase-associated lipocalin (NGAL) and HA. In addition, the metabolic biochemical parameters were also investigated. These parameters included levels of sodium, potassium, calcium, magnesium, ammonia, phosphate, sulphate, oxalate, citrate, urate, chloride and creatinine.The pH and osmolality were also investigated.

The preliminary results have confirmed that urinary HA is a reliable indicator of active or silent stones. The investigators reported this earlier in the initial findings of the presence of urinary HA. The proportion of excreted HA was significantly high. This finding was reported at the October 2018 meeting of the Société Internationale d'Urologie held in Seoul, Korea. HA is a ubiquitously distributed component of the extracellular matrix. In its native form, it exists as a high-molecular weight polymer, and lower-molecular weight forms of HA species accumulate at sites of inflammation and tissue injury. Previous studies concur that urinary HA is composed predominantly of lower-molecular weight (~10 kDa) species , which suggests a role for these species as mediators of inflammation.

Of the inflammatory and urinary biochemical markers, IL-6 and IL-8 were predictably higher, and NGAL was also significantly increased compared to controls and patients who had stones removed. It is also interesting to note that the stone-former cohorts had lower citrate and higher oxalate excretion, although just at the trend level. However, the medians differed clearly from those of the control group, suggesting that the measurement of citrate and oxalate is still a useful indicator of the risk of stone formation.

Therefore in this follow-up study, the investigators would like to investigate the time points at which recurrent stone-formers should be monitored over the longitudinal study period proposed herein.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Chinese male patients with age > 18 years old
2. History of radio-opaque urinary calculi with treatment performed (including spontaneous passage) and now stone free.

Exclusion Criteria:

* Patient refused or unable to provide consent for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with history of radio-opaque urinary calculi with treatment performed (including spontaneous passage) and now stone free.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Investigate the time points at which recurrent stone-formers should be monitored over the longitudinal study period and relate biomarker changes to clinical signs and data. | up to 24 months
  Patient will be reviewed with early morning urine collection for a complete urinalysis and biomarkers measurement every three months. The inflammatory cytokine expression of RNA retrieved from patient urine will be assessed. There will be radiological testing to check if there is any suspect stone.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong